CLINICAL TRIAL: NCT04231084
Title: Acute Hemodynamic Comparison of Inhaled Nitric Oxide and Inhaled Epoprostenol in Pulmonary Hypertension
Brief Title: Comparison of Vasodilator Response of Inhaled Epoprostenol and Inhaled Nitric Oxide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Aaron Waxman MD PhD, Associate Professor of Pulmonary and Critical Care, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2019P003491
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2023-02

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled Nitric Oxide (Active Comparator): Vasodilator testing will be performed with inhaled nitric oxide
  Interventions: Drug: Vasodilator testing (Inhaled Nitric Oxide)
- Inhaled Epoprostenol (Experimental): Vasodilator testing will be performed with inhaled epoprostenol
  Interventions: Drug: Vasodilator testing (Inhaled Epoprostenol)

INTERVENTIONS:
Drug: Vasodilator testing (Inhaled Nitric Oxide) — Right heart catheterization with vasodilator testing with each arms' associated agent will be performed
  Arms: Inhaled Nitric Oxide
Drug: Vasodilator testing (Inhaled Epoprostenol) — Right heart catheterization with vasodilator testing with each arms' associated agent will be performed
  Arms: Inhaled Epoprostenol

SUMMARY:
The overarching goal of this study is to examine the acute vasoreactive response to both inhaled nitric oxide and inhaled epoprostenol across both traditionally and non-traditionally interrogated phenotypes in PH, and to further characterize the relationship of vasoreactivity to disease severity and PH phenotype.

ELIGIBILITY:
Inclusion Criteria:

* mPAP ≥ 21mmHg, PAWP ≤ 25mmHg, and PVR ≥3 WU
* Classified as WHO group I-III pulmonary hypertension

Exclusion Criteria:

* WHO group IV and V pulmonary hypertension
* Patients who are on baseline pulmonary vasodilator medications
* Severe aortic or mitral valve disease
* Patients who are pregnant
* Left ventricular ejection fraction of <35%
* Patients who are hospitalized as inpatients at the time of RHC
* Patients with systolic blood pressure <90mmHg or mean arterial pressure of < 60mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in mean pulmonary artery pressure | Pre-pulmonary vasodilator testing measurements (baseline) will be compared to post-pulmonary vasodilator testing measurements during diagnostic right heart catheterization.
  The primary outcome will be change in mean pulmonary artery pressure (mmHg) from baseline to after 5-minutes of inhaled vasodilator.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron B Waxman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once study completion achieved